CLINICAL TRIAL: NCT01448720
Title: Treatment of Patients With Recently Exacerbated Schizophrenia With Paliperidone Palmitate - A Pilot Study
Brief Title: Treatment of Patients With Recently Exacerbated Schizophrenia With Paliperidone Palmitate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017977; R092670SCH3012 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2011-09-06; First posted 2011-10-07 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone palmitate; Long-acting injectable antipsychotic medication
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone palmitate (Experimental)
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — Type=exact number, unit=mg, number=150, 100, 75 mg equivalent (eq), form=suspension for injection, route=intramuscular use. One IM injection of 150 mq on Day 1, 100 mg eq. on Day 8 (+/- 4 days), and 75 mg eq. is recommended on Days 36, 64, and 92.

SUMMARY:
The purpose of this study is to explore the efficacy of paliperidone palmitate administered as a once monthly injection in patients with an acute exacerbation of schizophrenia.

DETAILED DESCRIPTION:
This is an open-label (patients and study staff will know the identity of treatments assigned) study of paliperidone palmitate in patients with acute an exacerbation of schizophrenia. The total duration of the study will be approximately 4 months. Eligible patients without a documented history of exposure to oral risperidone or paliperidone extended-release (ER), or intramuscular (IM) RISPERDAL CONSTA or paliperidone palmitate will receive oral risperidone 1 mg/day or extended release (ER) OROS paliperidone 3 mg/day for at least 3 days before the first injection of the study drug (paliperidone palmitate) for tolerability testing. Paliperidone palmitate will be administered to patients as an intramuscular (IM) injection in the deltoid (upper arm) or gluteal (buttocks) muscle.

ELIGIBILITY:
Inclusion Criteria:

* Be otherwise healthy on the basis of physical examination and vital signs at Screening (Baseline) and have a current diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) for at least 1 year before screening and no longer than 5 years (early diagnosed patients)
* Have acute exacerbation of psychosis defined as: less than 4 weeks but more than 4 days, PANSS total score of 70 to 120 (inclusive) at screening (moderate symptomatology), a score of 4 or more (at least moderately ill) at screening on the severity scale of the CGI-S
* If a woman, before entry she must be postmenopausal for at least 1 year, surgically sterile or abstinent. If sexually active, agree to practice an effective method of birth control before entry and throughout the study as specified in the protocol; If a man is heterosexually active with a woman of childbearing potential, he must agree to use a double-barrier method of birth control and to not donate sperm during the study and for 50 days after receiving the last dose of the study drug

Exclusion Criteria:

* Has evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal, neurological, endocrine, metabolic or pulmonary disease in the past 6 months (as determined by medical history, clinical laboratory or electrocardiogram [ECG] results, or physical examination) that would increase the risk associated with taking study medication or would confound the interpretation of the study
* The psychiatric diagnosis is due to direct pharmacological effects of a substance (eg, a drug of abuse or medication) or a general medical condition (eg, clinically notable hypothyroidism, delirium)
* Meets the DSM-IV definition of substance dependence (except for nicotine and caffeine) within 6 months prior to entry
* Has history or current symptoms of tardive dyskinesia (involuntary repetitive body movements)
* Has history of neuroleptic malignant syndrome

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in the Positive and Negative Syndrome Scale (PANSS) | Baseline to 4 months
  The neuropsychiatric symptoms of schizophrenia will be assessed using the 30-item PANSS, which provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items). Each question is rated on a scale of 1 (absent) to 7 (extreme).

SECONDARY OUTCOMES:
Change from Baseline in global severity of illness using the clinical global impression - severity (CGI-S) scores | Baseline to 4 months
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, the patient will be assessed on severity of mental illness at the time of rating between 1 (not ill) and 7 (extremely severe).
Change from Baseline in the personal and social performance scale (PSP) | Baseline to 4 months
  The PSP scale assesses the degree of dysfunction a patient exhibits over a 7-day period within 4 domains of behavior:(a) socially useful activities, (b) personal and social relationships, (c) self-care, and (d) disturbing and aggressive behavior. A score between 71 and 100 indicates only mild difficulties, and one between 31 and 70 indicates varying degrees of disability. A patient with a score of 30 or less has functioning so poor he or she requires intensive support or supervision..

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (12):
- Brazil (4):
  - Porto Alegre
  - Riberao Preto
  - São José
  - São Paulo
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Bucarmanga
  - Medellín
- Mexico (4):
  - Acapulco
  - Guadalajara
  - México
  - Monterrey

REFERENCES:
- See also: Treatment of Patients With Recently Exacerbated Schizophrenia With Paliperidone Palmitate - A Pilot Study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2510&filename=CR017977_CSR.pdf